CLINICAL TRIAL: NCT06790524
Title: Evaluation of Peri-implant Bone Changes Around One-piece Implant and Two-piece Implants Supporting Mandibular Screw-retained All-On-Four Full Arch Prosthesis: a Randomized Controlled Clinical Trial
Brief Title: Comparative Evaluation Between One-piece and Two-piece Implants Supporting Mandibular Screw-retained All-On-Four Full-arch Prosthesis on Peri-implant Bone Changes.
Acronym: RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Khaled Hassan Mahdy, Master degree candidate at Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: one-piece implants
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-01

CONDITIONS: Marginal Bone Loss; One-piece Implants Versus Two-piece Implants During the Osseointegration Phase
Keywords: one-piece implants , All-On-Four, Marginal bone loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients will receive an implant screw-retained restoration supported by One-piece implants. (Experimental): One-piece dental implants with multi-unit abutments mounted on them, provided with different implant-abutment angulation which makes them utilizable for All-On-Four prosthesis.
  Interventions: Device: One-piece dental implants with MUA
- Patients will receive an implant screw-retained restoration supported by two-piece implants. (Active Comparator): Two-piece Implants, Implant fixtures, and separate pieces of Multi-unit abutments with different angulations will be used to support the All-On-Four prostheiss.
  Interventions: Device: Two-piece dental implants

INTERVENTIONS:
Device: One-piece dental implants with MUA — one-piece dental implants with multi-units abutment mounted on the implants as a single piece provided with different abutment angulation utilizing these implants for All-On-Four prothesis
  Other Names: single piece implants; mono implenats
  Arms: Patients will receive an implant screw-retained restoration supported by One-piece implants.
Device: Two-piece dental implants — Surgical and immediate loading procedures:
  On the day of implant placement, patients will receive two-piece implant. After crestal incision and full-thickness flap elevation, the implant sites will be prepared aided by a surgical template. 4 implants will be placed, two aligned in an axial orientation and two will be distally aligned (17 degrees). The standard placement procedure as recommended by the manufacturer will be used. The surgical drills with increasing diameters will be used to prepare the implant sites. Implants will be ideally placed at bone level (or 1 mm deeper depending on the soft tissue thickness). After 3 months as a healing phase, a definitive prosthesis will be fabricated using the same abutments, and the marginal bone loss after the osseointegration phase will be assessed.
  Other Names: endosteal implants; root form implants
  Arms: Patients will receive an implant screw-retained restoration supported by two-piece implants.

SUMMARY:
Evaluating the bone changing after receiving one-piece implants supported full arch prosthesis compared to the conventional two-piece implants.

DETAILED DESCRIPTION:
Studying the difference between one-piece and two-piece implants and their effect on bone loss. This will help in simplifying the surgical procedure for full arch implant-supported prosthesis rehabilitation using one-piece implants, eliminating the disturbance of the gum tissue around the implants, potentially reducing the risk of bacterial colonization and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients, who can sign an informed consent will be considered eligible for this trial.
* Residual bone height should have sufficient volume and quality for implant placement with a minimum of 12-14 mm in height and 6 mm in width.
* Patients who already have existing maxillary and mandibular complete dentures, and after examination of the mandibular dentures, technical problems concerning denture design and/or occlusion are found, or who are dissatisfied with the retention and stability of their technically satisfactory mandibular dentures.

Exclusion Criteria:

* - Patients with conditions that may contraindicate implant placement (e.g., Immunosuppressed or immunocompromised patients, patients under treatment of intravenous amino bisphosphonates, patients undergoing radiotherapy to the head and neck region).
* Inadequate mouth opening
* Heavy smokers, more than 10 cigarettes/day
* Patients with poor oral hygiene and motivation.
* Pregnancy or nursing.
* Drug abusers.
* Psychiatric problems or unrealistic expectations.
* Patients with infection and or inflammation in the area intended for implant placement.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Peri-implant marginal bone loss | From implant placement (baseline) and After 3 months (after the osseointegration phase)
  Peri-implant marginal bone loss will be assessed utilizing CBCT. The radiographic evaluation will be performed at baseline and at 3 months after functional loading. Using the first thread of the implant as a standard reference point, the circumference of the Crestal bone level around the implant will be measured in all directions (mesial, distal, buccal, and lingual) in width and height.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No